CLINICAL TRIAL: NCT06472440
Title: Evaluation of the Use of a Method "Radiomics" for Positons Emission Tomography With Fluor-18-Fluoro-DOPA PET in Gliomas
Brief Title: Evaluation of the Use of a Method "Radiomics" for DOPA PET in Gliomas
Acronym: RADDOPAG-2
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Professor of University and Medical Doctor, MD PhD, Central Hospital, Nancy, France
Other Study IDs: 2024PI089
Record Dates: First submitted 2024-05-17; First posted 2024-06-25 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
: The evaluation of gliomas in imaging represents a real challenge today, at the initial diagnosis, for therapeutic planning or follow-up treatment of these lesions. There is an urgent need for non-invasive imaging tools to evaluate a glioma throughout its management. At present, the diagnosis of certainty is only obtained through an anatomo-pathological analysis with sampling during an invasive procedure (surgery or biopsy). Magnetic resonance imaging, through perfusion, diffusion imaging or spectroscopy is developing in gliomas. However, it remains time-consuming and is not always available. At the same time, positron emission tomography (PET) with amino acids is an interesting alternative for these brain tumours. Amino acid PET has the advantage of being more specific than the abnormalities detected in MRI and the amino acid radiotracers cross the blood-brain barrier, even if not broken, unlike Gadolinium in MRI. Among these radiotracers, 18F-FDOPA can, among other things, assist in the non-invasive staging of gliomas at initial diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Patient having performed a PET/CT examination at 18F-FDOPA for his glioma in the nuclear medicine department of the CHRU de Brabois for which the raw data are available;
* Person who received full information on the organization of the research and did not object to the use of these data;
* Patients affiliated to a social security scheme

Exclusion Criteria:

Person who received full information on the organization of the research and who objected to the use of the data

* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice).
* A person of full age who is unable to give consent and who is not subject to a legal protection measure.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a brain PET/CT examination using 18F-FDOPA (between 01/JAN/2020 and 01/JUN/2024) and presenting a histologically confirmed glioma
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-11-16 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance (sensitivity, specificity, accuracy) of parameters extracted from radiomic analysis to predict the molecular characteristics of gliomas at initial diagnosis. | Day 1
  Accuracy of the method

SECONDARY OUTCOMES:
Diagnostic performance (sensitivity, specificity, accuracy) of parameters extracted from radiomic analysis to predict glioma recurrence | Day 1
  Sensibility of the method
Diagnostic performance (sensitivity, specificity, accuracy) of parameters extracted from radiomic analysis to predict the response to glioma treatments. | Day 1
  specificity of the method

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of NANCY, Vandœuvre-lès-Nancy, France